CLINICAL TRIAL: NCT05707962
Title: A Multicentre Double Blind Trial of the Neuroprotective Efficacy of Postnatal Magnesium Sulphate in Term/Near Term Infants With Moderate to Severe Birth Asphyxia
Brief Title: Neuroprotective Efficacy of Postnatal Magnesium Sulphate in Term Infants With Birth Asphyxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Komal Khadim Hussain, principal investigator, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB/2022/1018/SIMS
Record Dates: First submitted 2023-01-22; First posted 2023-02-01 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Birth Asphyxia
Keywords: birth asphyxia; magnesium sulphate; term infants
MeSH Terms: conditions — Asphyxia Neonatorum | interventions — Magnesium Sulfate; Neuroprotective Agents

STUDY DESIGN:
Intervention Model Description: All babies with moderate or severe Hypoxic Ischemic Encephalopathy fulfilling the inclusion criteria will be randomized to receive either the standard treatment (oxygen and fluid therapy along with anticonvulsants if required) plus 3.0 ml/kg of 10% dextrose water given over 30 minutes, three dose given 24 hours apart or to receive standard treatment PLUS three doses of Magnesium Sulphate infusion given over 30 minutes at 250 mg/kg per dose given 24 hours apart. The volume of infusion shall be adjusted with 10% dextrose water to make it
Who Masked: Participant, Care Provider
Masking Description: As soon as parental consent has been obtained the baby will be allocated to one arm of the study using randomly shuffled sealed brown envelopes containing the allocation arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental): All babies with moderate or severe Hypoxic Ischemic Encephalopathy fulfilling the inclusion criteria will be randomized to receive either the standard treatment (oxygen and fluid therapy along with anticonvulsants if required) plus 3.0 ml/kg of 10% dextrose water given over 30 minutes, three dose given 24 hours apart or to receive standard treatment PLUS three doses of Magnesium Sulphate infusion given over 30 minutes at 250 mg/kg per dose given 24 hours apart. The volume of infusion shall be adjusted with 10% dextrose water to make it
  up to 3.0 ml. The resulting reconstituted solution for intravenous infusion shall be 8.3% Magnesium Sulphate delivered over 30 minutes at a rate of 0.1 ml/kg/minute i.e. 8.3 mg/kg/minute. The treatment should be started as soon after birth as possible and not later than 24 hours of life. The babies who meet the exclusion criteria will not be continued into the study.
  Interventions: Drug: Magnesium sulfate
- non intervention group (No Intervention): All babies with moderate or severe Hypoxic Ischemic Encephalopathy fulfilling the inclusion criteria will be randomized to receive either the standard treatment (oxygen and fluid therapy along with anticonvulsants if required) plus 3.0 ml/kg of 10% dextrose water given over 30 minutes, three dose given 24 hours apart or to receive standard treatment PLUS three doses of Magnesium Sulphate infusion given over 30 minutes at 250 mg/kg per dose given 24 hours apart. The volume of infusion shall be adjusted with 10% dextrose water to make it
  up to 3.0 ml. The resulting reconstituted solution for intravenous infusion shall be 8.3% Magnesium Sulphate delivered over 30 minutes at a rate of 0.1 ml/kg/minute i.e. 8.3 mg/kg/minute. The treatment should be started as soon after birth as possible and not later than 24 hours of life. The babies who meet the exclusion criteria will not be continued into the study.

INTERVENTIONS:
Drug: Magnesium sulfate — All babies with moderate or severe Hypoxic Ischemic Encephalopathy fulfilling the inclusion criteria will be randomized to receive either the standard treatment (oxygen and fluid therapy along with anticonvulsants if required) plus 3.0 ml/kg of 10% dextrose water given over 30 minutes, three dose given 24 hours apart or to receive standard treatment PLUS three doses of Magnesium Sulphate infusion given over 30 minutes at 250 mg/kg per dose given 24 hours apart. The volume of infusion shall be adjusted with 10% dextrose water to make it
  up to 3.0 ml. The resulting reconstituted solution for intravenous infusion shall be 8.3% Magnesium Sulphate delivered over 30 minutes at a rate of 0.1 ml/kg/minute i.e. 8.3 mg/kg/minute. The treatment should be started as soon after birth as possible and not later than 24 hours of life. The babies who meet the exclusion criteria will not be continued into the study.
  Other Names: neuroprotective agent
  Arms: intervention group

SUMMARY:
Birth/Perinatal asphyxia in Pakistan continues to be a leading cause of neonatal mortality and morbidity. It is estimated that around 80 to 120,000 neonates either suffer from or die from birth/perinatal asphyxia every year. In addition to the large number of deaths a larger number of babies who survive suffer from neuro-developmental disorders adding to the health burden to the society and the nation.

To date other than prevention (which requires global efforts to improve maternal education and health care) the therapies available to treat infants who have suffered from birth asphyxia have been either technically too complex or extremely expensive.

DETAILED DESCRIPTION:
Birth/Perinatal asphyxia in Pakistan continues to be a leading cause of neonatal mortality and morbidity. It is estimated that around 80 to 120,000 neonates either suffer from or die from birth/perinatal asphyxia every year. In addition to the large number of deaths a larger number of babies who survive suffer from neuro-developmental disorders adding to the health burden to the society and the nation.

To date other than prevention (which requires global efforts to improve maternal education and health care) the therapies available to treat infants who have suffered from birth asphyxia have been either technically too complex or extremely expensive.

Recent evidence from animal studies and small human studies it has become clear that giving Magnesium Sulphate to term or nearterm babies with moderate to severe birth/perinatal asphyxia reduces both mortality and morbidity.

Magnesium Sulphate as a drug has been in clinical use for decades; its pharmacokinetics, safety profile and mode of action are well known. It is cheap and readily available in Pakistan thus providing an opportunity to confirm or refute the efficacy of Magnesium Sulphate in birth/perinatal asphyxia.

With this in mind the following pragmatic study has been designed using the current practices and available resources:

ELIGIBILITY:
Inclusion Criteria:

* Term and near term infants (≥35 weeks gestation) with moderate to severe birth asphyxia Age at admission < 24 hours

Exclusion Criteria:

* Babies who could not be given first injection before 24 hours of age

Infants with major congenital malformations, sepsis, congenital heart defects, Intracranial hemorrhage and surgical problems

Babies received intubated in emergency

Babies receiving therapeutic hypothermia

Infants with disorders of metabolism

Infants in whom cause other than asphyxia is established as the reason for not initiating or sustaining breathing at birth.

Ages: 1 Hour to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 178 (Actual)
Dates: Start 2023-03-24 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
number of participants died (receiving mgso4) | 6 hours
  Mortality between the two groups (Standard management vs Magnesium Sulphate treated group). Further analyzed by the stage of asphyxia
number of participants diednumber (difference in time of administration) | 24 hours
  Mortality between the two groups (Standard management vs Magnesium Sulphate treated group) in those where magnesium sulphate was given within six hours of birth and those given later than six hours of birth.

SECONDARY OUTCOMES:
number of seizure episode | 6 hours
  Frequency of seizures in the two groups and number of days to achieve seizure control.
days in achieving full enteral feed | 1 month
  Number of days to achieve oral feed.
assessment of neurodevelopmental damage | 1 month
  Neurodevelopmental disability in survivors at 18 months of age as assessed by a developmental pediatrician blinded to the study groups using one standard developmental screening method in all babies

CONTACTS AND LOCATIONS:
Overall Officials: dr sikandar hayat, MBBS, FCPS, Study Chair — children hospital Lahore
Locations (1):
- services hospital Pakistan, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data will be collected on data record forms (DRFs) given in appendix 1. Short-term outcomes include initiation of feed in days, seizure control in days, duration of stay, cranial ultrasound findings and EEG at discharge or last reported before death and discharge or death will be recorded. Cranial ultrasound and EEG will be performed by the same sonologist and neurologist. The developmental assessment will be done at 18 months of age by the same neurodevelopmental pediatrician, blinded to the study using Griffiths scoring system.